CLINICAL TRIAL: NCT01454739
Title: An Open-Label, Multicenter Evaluation of the Long-Term Safety and Efficacy of Recombinant Human Coagulation Factor VIII Fusion Protein (rFVIIIFc) in the Prevention and Treatment of Bleeding Episodes in Previously Treated Subjects With Hemophilia A
Brief Title: Long-Term Safety and Efficacy of rFVIIIFc in the Prevention and Treatment of Bleeding Episodes in Previously Treated Participants With Hemophilia A
Acronym: ASPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioverativ Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8HA01EXT; 2011-003072-37
Record Dates: First submitted 2011-09-29; First posted 2011-10-19 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2018-11

CONDITIONS: Hemophilia A
Keywords: rFVIIIFc; A-LONG Extension
MeSH Terms: conditions — Hemophilia A | interventions — factor VIII-Fc fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- On-Demand (Experimental): The individual dose of rFVIIIFc to treat bleeding episodes will be based on participant's clinical condition, type and severity of the bleeding event, and if indicated, Factor VIII (FVIII) levels.
  Interventions: Drug: rFVIIIFc
- Prophylaxis (Experimental): Tailored prophylaxis, Weekly prophylaxis or Personalized prophylaxis available.
  Interventions: Drug: rFVIIIFc

INTERVENTIONS:
Drug: rFVIIIFc — Administered as specified in the treatment arm.
  Other Names: Eloctate; recombinant coagulation factor VIII Fc fusion protein; BIIB031; antihemophilic factor (recombinant) Fc fusion protein; efmoroctocog alfa

SUMMARY:
The primary objective of the study is to evaluate the long-term safety of recombinant human Factor VIII Fc fusion protein (rFVIIIFc) in participants with hemophilia A. The secondary objective of the study is to evaluate the efficacy of rFVIIIFc in the prevention and treatment of bleeding episodes in participants with hemophilia A.

DETAILED DESCRIPTION:
Participant will follow either a prophylaxis or on-demand regimen. The starting dose in this study will be determined by the clinical profile of the participant in the preceding studies A-LONG - 997HA301 (NCT01181128), pediatric study 8HA02PED (NCT01458106), 997HA307 (NCT02083965) and 997HA309 (NCT02502149).

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects who have completed previous rFVIIIFc studies (NCT01181128, NCT02083965, NCT01458106 and NCT02502149)
* Ability to understand purposes and risks of the study and to provide signed and dated informed consent (or assent, as applicable).

Key Exclusion Criteria:

* Confirmed positive high-titer inhibitor (≥5.00 BU/mL).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 0 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Bioverativ Therapeutics Inc.
Locations (73):
- United States (20):
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Indianapolis, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, New Orleans, Louisiana
  - Research Site, Boston, Massachusetts
  - Research Site, East Lansing, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington
- Australia (7):
  - Research Site, Camperdown, New South Wales
  - Research Site, South Brisbane, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Melbourne, Victoria
  - Research site, Melbourne, Victoria
  - Research Site, Murdoch, Western Australia
  - Research Site, Subiaco, Western Australia
- Research Site, Vienna, Austria
- Research Site, Brussels, Brussels Capital, Belgium
- Research Site, Campinas, São Paulo, Brazil
- Canada (2):
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
- Research Site, Bron, Rhone, France
- Germany (2):
  - Research Site, Bonn, North Rhine-Westphalia
  - Research Site, Berlin
- Hong Kong (3):
  - Children Cancer Centre, Hong Kong, New Territories
  - Sir Yue Kong Pao Center for Cancer, Hong Kong, New Territories
  - Research Site, Hong Kong
- India (5):
  - Research Site, Bangalore, Karnataka
  - Research Site, Pune, Maharashtra
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Ludhiana, Punjab
  - Research Site, Vellore, Tamil Nadu
- Research Site, Dublin, Ireland
- Research Site, Ramat Gan, Israel
- Italy (3):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Vicenza
- Japan (6):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Kitakyushu, Fukuoka
  - Research Site, Kawasaki, Kanagawa
  - Research Site, Kashihara-shi, Nara
  - Research Site, Shinjuku-ku, Tokyo-To
  - Research Site, Tokyo, Tokyo-To
- Research Site, Groningen, Netherlands
- New Zealand (5):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research site, Hamilton
  - Research Site, Palmerston North
  - Research site, Wellington
- Research Site, Lublin, Poland
- South Africa (2):
  - Research Site, Johannesburg, Gauteng
  - Research Site, Cape Town, Western Cape
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- Research Site, Gothenburg, Sweden
- Research Site, Zurich, Switzerland
- United Kingdom (6):
  - Research Site, Cambridge, Cambridgeshire
  - Research Site, London, Greater London
  - Research Site, Basingstoke, Hampshire
  - Research Site, Hamstead, London
  - Research Site, Glasgow, Strathclyde
  - Research Site, London

REFERENCES:
- [Derived] Raheja P, Kragh N, Bystricka L, Eriksson D, Aroui K, Mezghani M, Barbier S, Linari S. Long-term efmoroctocog alfa prophylaxis improves perceived pain, mental, and physical health in patients with hemophilia A: post hoc analysis of phase III trials using patient-reported outcomes. Ther Adv Hematol. 2024 Jul 30;15:20406207241257917. doi: 10.1177/20406207241257917. eCollection 2024. PMID 39091324
- [Derived] Nolan B, Mahlangu J, Pabinger I, Young G, Konkle BA, Barnes C, Nogami K, Santagostino E, Pasi KJ, Khoo L, Winding B, Yuan H, Fruebis J, Rudin D, Oldenburg J. Recombinant factor VIII Fc fusion protein for the treatment of severe haemophilia A: Final results from the ASPIRE extension study. Haemophilia. 2020 May;26(3):494-502. doi: 10.1111/hae.13953. Epub 2020 Mar 30. PMID 32227570
- [Derived] Nolan B, Mahlangu J, Perry D, Young G, Liesner R, Konkle B, Rangarajan S, Brown S, Hanabusa H, Pasi KJ, Pabinger I, Jackson S, Cristiano LM, Li X, Pierce GF, Allen G. Long-term safety and efficacy of recombinant factor VIII Fc fusion protein (rFVIIIFc) in subjects with haemophilia A. Haemophilia. 2016 Jan;22(1):72-80. doi: 10.1111/hae.12766. Epub 2015 Jul 27. PMID 26218032

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed studies 8HA02PED [NCT01458106], 997HA301 [NCT01181128]), 997HA307 (NCT02083965) and 997HA309 (NCT02502149) were expected to be eligible to enroll in this study.
Groups:
- rFVIIIFc (Participants From Study 8HA02PED): Participants received rFVIIIFc intravenously (IV) per assigned treatment regimen as follows: Tailored Prophylaxis(TP): 25 IU/kg-65 IU/kg rFVIIIFc every 3-5 days or 2 times/week at approximately 20 IU/kg to 65 IU/kg rFVIIIFc on Day 1 and 40 IU/kg-65 IU/kg rFVIIIFc on Day 4. Weekly P(WP): rFVIIIFc once weekly at approximately 65 IU/kg. Personalized P: If optimal prophylaxis dosing not achieved using TP/WP, Investigator personalized dosing to meet individual participant's needs (i.e. adding prevention dose prior to strenuous activity; targeting FVIII trough level of >3%, if bleeding history and/or activity level requires/dosing less frequently). Episodic (On demand): individual dose of rFVIIIFc based on clinical condition, type and severity of bleeding event and if indicated, FVIII levels (per investigator and Sponsor decision). For participants <12 years, weekly and episodic treatment regimens were only available once reached at age of 12 years old.
- rFVIIIFc(Participants From Studies 997HA301/997HA307/997HA309): Participants received rFVIIIFc IV as per their assigned treatment regimen as follows: Tailored Prophylaxis (TP): 25 international unit per kilogram (IU/kg)-65 IU/kg rFVIIIFc every 3-5 days or 2 times/week at approximately 20 IU/kg to 65 IU/kg rFVIIIFc on Day 1 and 40 IU/kg-65 IU/kg rFVIIIFc on Day 4. Weekly P: rFVIIIFc once weekly at approximately 65 IU/kg. Personalized P: If optimal prophylaxis dosing not achieved using TP/WP, Investigator personalized dosing to meet individual participant's needs (options: adding "prevention" dose prior to strenuous activity; targeting FVIII trough level of greater than (>)3 percent (%), if bleeding history and/or activity level requires/dosing less frequently. Episodic (On demand): individual dose of rFVIIIFc based on clinical condition, type and severity of bleeding event and if indicated, FVIII levels (per investigator and Sponsor decision). The rate of administration determined by participant's comfort level.
Period: Overall Study
Arm/Group | rFVIIIFc (Participants From Study 8HA02PED) | rFVIIIFc(Participants From Studies 997HA301/997HA307/997HA309)
Started | 61 (30 participants in <6 Years Old Age Cohort and 31 participants in 6 to <12 Years Old Age Cohort.) | 179
Tailored Prophylaxis | 59 | 131
Weekly Prophylaxis | 0 | 34
Personalized Prophylaxis | 3 | 23
Episodic | 0 | 13
Surgery Subgroup (Participants who have undergone major surgery or have major surgical/rehabilitation period in study.) | 2 | 26
Completed | 54 | 158
Not Completed | 7 | 21
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Other | 3 | 5
Not completed — Physician Decision | 0 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- rFVIIIFc (Participants From Study 8HA02PED): Participants received rFVIIIFc IV per assigned treatment regimen as follows: Tailored Prophylaxis(TP): 25 IU/kg-65 IU/kg rFVIIIFc every 3-5 days or 2 times/week at approximately 20 IU/kg to 65 IU/kg rFVIIIFc on Day 1 and 40 IU/kg-65 IU/kg rFVIIIFc on Day 4. Weekly P: rFVIIIFc once weekly at approximately 65 IU/kg. Personalized P: If optimal prophylaxis dosing not achieved using TP/WP, Investigator personalized dosing to meet individual participant's needs (i.e. adding "prevention" dose prior to strenuous activity; targeting FVIII trough level of >3%, if bleeding history and/or activity level requires/dosing less frequently). Episodic (On demand): individual dose of rFVIIIFc based on clinical condition, type and severity of bleeding event and if indicated, FVIII levels (per investigator and Sponsor decision). For participants less than (<)12 years of age, weekly and episodic treatment regimens were only available once reached at age of 12 years old.
- rFVIIIFc(Participants From Studies 997HA301/997HA307/997HA309): Participants received rFVIIIFc IV per assigned treatment regimen as follows: Tailored Prophylaxis (TP): 25 IU/kg-65 IU/kg rFVIIIFc every 3-5 days or 2 times/week at approximately 20 IU/kg to 65 IU/kg rFVIIIFc on Day 1 and 40 IU/kg-65 IU/kg rFVIIIFc on Day 4. Weekly P: rFVIIIFc once weekly at approximately 65 IU/kg. Personalized P: If optimal prophylaxis dosing not achieved using TP/WP, Investigator personalized dosing to meet individual participant's needs (options: adding "prevention" dose prior to strenuous activity; targeting FVIII trough level of greater than >3 %, if bleeding history and/or activity level requires/dosing less frequently. Episodic (On demand): individual dose of rFVIIIFc based on clinical condition, type and severity of bleeding event and if indicated, FVIII levels (per investigator and Sponsor decision). The rate of administration determined by participant's comfort level.
- Total: Total of all reporting groups
Arm/Group | rFVIIIFc (Participants From Study 8HA02PED) | rFVIIIFc(Participants From Studies 997HA301/997HA307/997HA309) | Total
Number analyzed (Participants) | 61 | 179 | 240
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 61 | 22 | 83
  Between 18 and 65 years | 0 | 156 | 156
  > 65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 61 | 179 | 240
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 8 | 10
  Not Hispanic or Latino | 59 | 147 | 206
  Unknown or Not Reported | 0 | 24 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 42 | 101 | 143
  Black or African American | 8 | 8 | 16
  Asian | 4 | 39 | 43
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Other | 7 | 7 | 14
  Unknown or Not Reported | 0 | 24 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Positive Inhibitor Development
Description: An inhibitor test result greater than or equal to (>=) 0.6 Bethesda units per milliliter (BU/mL), identified and confirmed by re-testing of a second sample obtained within 2 to 4 weeks, was considered positive. Both tests were to be performed using the Nijmegen-modified Bethesda Assay by the central laboratory. Data was summarized by treatment regimen for participants from 997HA301/997HA307/997HA309 combined and by age cohort (<6 years and 6 to <12 years old) and treatment regimen for participants from 8HA02PED per planned analysis. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Approximately 5 years
Population: Safety analysis set included participants who received at least 1 dose of Recombinant Human Coagulation Factor VIII Fusion Protein(rFVIIIFc) in study 8HA01EXT.
Measure: Count of Participants; unit: Participants
Groups:
- rFVIIIFc (8HA02PED [<6 Years Old Age Cohort]): Participants with < 6 years old age received rFVIIIFc IV per assigned treatment regimen as follows: Tailored Prophylaxis(TP): 25 IU/kg-65 IU/kg rFVIIIFc every 3-5 days or 2 times/week at approximately 20 IU/kg to 65 IU/kg rFVIIIFc on Day 1 and 40 IU/kg-65 IU/kg rFVIIIFc on Day 4. Weekly P: rFVIIIFc once weekly at approximately 65 IU/kg. Personalized P: If optimal prophylaxis dosing not achieved using TP/WP, Investigator personalized dosing to meet individual participant's needs (i.e. adding "prevention" dose prior to strenuous activity; targeting FVIII trough level of >3%, if bleeding history and/or activity level requires/dosing less frequently). Episodic (On demand): individual dose of rFVIIIFc based on clinical condition, type and severity of bleeding event and if indicated, FVIII levels (per investigator and Sponsor decision). For participants <12 years of age, weekly and episodic treatment regimens were only available once reached at age of 12 years old.
- rFVIIIFc (8HA02PED [6 to <12 Years Old Age Cohort]): Participants with 6 to <12 years old age received rFVIIIFc IV per assigned treatment regimen as follows: Tailored Prophylaxis(TP): 25 IU/kg-65 IU/kg rFVIIIFc every 3-5 days or 2 times/week at approximately 20 IU/kg to 65 IU/kg rFVIIIFc on Day 1 and 40 IU/kg-65 IU/kg rFVIIIFc on Day 4. Weekly P: rFVIIIFc once weekly at approximately 65 IU/kg. Personalized P: If optimal prophylaxis dosing not achieved using TP/WP, Investigator personalized dosing to meet individual participant's needs (i.e. adding "prevention" dose prior to strenuous activity; targeting FVIII trough level of >3%, if bleeding history and/or activity level requires/dosing less frequently). Episodic (On demand): individual dose of rFVIIIFc based on clinical condition, type and severity of bleeding event and if indicated, FVIII levels (per investigator and Sponsor decision). For participants <12 years of age, weekly and episodic treatment regimens were only available once reached at age of 12 years old.
Arm/Group | rFVIIIFc (8HA02PED [<6 Years Old Age Cohort]) | rFVIIIFc (8HA02PED [6 to <12 Years Old Age Cohort]) | rFVIIIFc(Participants From Studies 997HA301/997HA307/997HA309)
Number analyzed (Participants) | 30 | 31 | 179
Participants | 0 | 0 | 0

2. Secondary Outcome: Annualized Bleeding Rate (ABR)
Description: ABR is annualized number of bleeding episodes per participant per year. Bleeding episodes were classified as spontaneous if participant records bleeding event when there is no known contributing factor such as definite trauma/antecedent strenuous activity and as traumatic if participant records bleeding event when there is known reason for bleed. ABR=(Number of bleeding episodes during efficacy period (EP)/number of days during EP)*365.25. EP reflects sum of all intervals of time during which participants were treated with rFVIIIFc per treatment regimen excluding major and minor surgical/rehabilitation periods and large injection intervals. ABR was summarized by treatment regimen for participants from studies 997HA301/997HA307/997HA309 combined and by age cohort (<6 years and 6 to <12 years old) and treatment regimen for participants from Study 8HA02PED per planned analysis. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Approximately 5 years
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of rFVIIIFc. Here 'n' (number analyzed) signifies number of participants who were analyzed in each treatment regimen, for each arm, respectively.
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | rFVIIIFc (8HA02PED [<6 Years Old Age Cohort]) | rFVIIIFc (8HA02PED [6 to <12 Years Old Age Cohort]) | rFVIIIFc(Participants From Studies 997HA301/997HA307/997HA309)
Number analyzed (Participants) | 30 | 31 | 179
episodes per participant per year
  Tailored Prophylaxis: number analyzed (Participants) | 29 | 30 | 131
  Tailored Prophylaxis | 1.18 [0.60 to 2.37] | 1.59 [0.55 to 3.55] | 0.64 [0.00 to 2.84]
  Weekly Prophylaxis: number analyzed (Participants) | 0 | 0 | 34
  Weekly Prophylaxis |  |  | 1.90 [0.27 to 4.85]
  Personalized Prophylaxis: number analyzed (Participants) | 2 | 1 | 23
  Personalized Prophylaxis | 3.72 [3.35 to 4.09] | 1.01 [1.01 to 1.01] | 4.11 [0.64 to 8.78]
  Episodic: number analyzed (Participants) | 0 | 0 | 13
  Episodic |  |  | 19.10 [15.12 to 30.46]

3. Secondary Outcome: Annualized Spontaneous Joint Bleeding Episodes
Description: Bleeding episodes were classified as spontaneous if participant records a bleeding event when there is no known contributing factor such as definite trauma/antecedent strenuous activity. In addition, location of bleed (joint, internal, skin/mucosa or muscle) were collected. Annualized spontaneous joint bleeding episodes=(Number of spontaneous joint bleeding episodes during efficacy period (EP)/number of days during EP)*365.25. EP reflects sum of all intervals of time during which participants were treated with rFVIIIFc per treatment regimen excluding major and minor surgical/rehabilitation periods and large injection intervals. Bleeding episodes were summarized by treatment regimen for participants from studies 997HA301/997HA307/997HA309 combined and by age cohort (<6 years and 6 to <12 years old) and treatment regimen for participants from Study 8HA02PED per planned analysis. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Approximately 5 years
Population: FAS included all participants who received at least 1 dose of rFVIIIFc. Here 'n' (number analyzed) signifies number of participants who were analyzed in each treatment regimen, for each arm, respectively.
Measure: Median (Inter-Quartile Range); unit: episodes per participant per year
Arm/Group | rFVIIIFc (8HA02PED [<6 Years Old Age Cohort]) | rFVIIIFc (8HA02PED [6 to <12 Years Old Age Cohort]) | rFVIIIFc(Participants From Studies 997HA301/997HA307/997HA309)
Number analyzed (Participants) | 30 | 31 | 179
episodes per participant per year
  Tailored Prophylaxis: number analyzed (Participants) | 29 | 30 | 131
  Tailored Prophylaxis | 0.00 [0.00 to 0.55] | 0.00 [0.00 to 0.55] | 0.00 [0.00 to 0.63]
  Weekly Prophylaxis: number analyzed (Participants) | 0 | 0 | 34
  Weekly Prophylaxis |  |  | 0.58 [0.00 to 1.90]
  Personalized Prophylaxis: number analyzed (Participants) | 2 | 1 | 23
  Personalized Prophylaxis | 2.20 [1.34 to 3.07] | 0.00 [0.00 to 0.00] | 0.91 [0.00 to 2.84]
  Episodic: number analyzed (Participants) | 0 | 0 | 13
  Episodic |  |  | 9.22 [4.35 to 15.70]

4. Secondary Outcome: Total Number of Exposure Days (EDs)
Description: An exposure day is a 24-hour period in which one or more rFVIIIFc injections are given. The total number of days of exposure to rFVIIIFc were summarized by treatment regimen for participants from studies 997HA301/997HA307/997HA309 combined and by age cohort (<6 years and 6 to <12 years old) and treatment regimen for participants from Study 8HA02PED per planned analysis. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Approximately 5 years
Population: Safety Analysis Set included participants who received at least 1 dose of rFVIIIFc in study 8HA01EXT. Here 'n' (number analyzed) signifies number of participants who were analyzed in each treatment regimen, for each arm, respectively.
Measure: Median (Full Range); unit: days
Arm/Group | rFVIIIFc (8HA02PED [<6 Years Old Age Cohort]) | rFVIIIFc (8HA02PED [6 to <12 Years Old Age Cohort]) | rFVIIIFc(Participants From Studies 997HA301/997HA307/997HA309)
Number analyzed (Participants) | 30 | 31 | 179
days
  Tailored Prophylaxis: number analyzed (Participants) | 29 | 30 | 131
  Tailored Prophylaxis | 287.00 [18.0 to 447.0] | 373.00 [85.0 to 467.0] | 257.00 [4.0 to 660.0]
  Weekly Prophylaxis: number analyzed (Participants) | 0 | 0 | 34
  Weekly Prophylaxis |  |  | 203.50 [5.0 to 318.0]
  Personalized Prophylaxis: number analyzed (Participants) | 2 | 1 | 23
  Personalized Prophylaxis | 127.00 [102.0 to 152.0] | 107.0 [107.0 to 107.0] | 223.00 [14.0 to 535.0]
  Episodic: number analyzed (Participants) | 0 | 0 | 13
  Episodic |  |  | 27.00 [0.0 to 88.0]

5. Secondary Outcome: Annualized rFVIIIFc Consumption (International Units Per Kilogram [IU/kg])
Description: Annualized consumption = (total international unit per kilogram [IU/kg] of study treatment received during the efficacy period / total number of days during the efficacy period) multiplied by 365.25. Efficacy period reflects sum of all intervals of time during which participants were treated with rFVIIIFc per treatment regimen excluding major and minor surgical/rehabilitation periods and large injection intervals. Annualized consumption was summarized by treatment regimen for participants from studies 997HA301/997HA307/997HA309 combined and by age cohort (<6 years and 6 to <12 years old) and treatment regimen for participants from Study 8HA02PED per planned analysis. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Time Frame: Approximately 5 years
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: IU per kilogram per year
Groups:
- rFVIIIFc[Participants From Studies 997HA301/997HA307/997HA309]: Participants received rFVIIIFc IV per assigned treatment regimen as follows: Tailored Prophylaxis (TP): 25 IU/kg-65 IU/kg rFVIIIFc every 3-5 days or 2 times/week at approximately 20 IU/kg to 65 IU/kg rFVIIIFc on Day 1 and 40 IU/kg-65 IU/kg rFVIIIFc on Day 4. Weekly P: rFVIIIFc once weekly at approximately 65 IU/kg. Personalized P: If optimal prophylaxis dosing not achieved using TP/WP, Investigator personalized dosing to meet individual participant's needs (options: adding "prevention" dose prior to strenuous activity; targeting FVIII trough level of greater than >3 %, if bleeding history and/or activity level requires/dosing less frequently. Episodic (On demand): individual dose of rFVIIIFc based on clinical condition, type and severity of bleeding event and if indicated, FVIII levels (per investigator and Sponsor decision). The rate of administration determined by participant's comfort level.
Arm/Group | rFVIIIFc (8HA02PED [<6 Years Old Age Cohort]) | rFVIIIFc (8HA02PED [6 to <12 Years Old Age Cohort]) | rFVIIIFc[Participants From Studies 997HA301/997HA307/997HA309]
Number analyzed (Participants) | 30 | 31 | 179
IU per kilogram per year
  Tailored Prophylaxis: number analyzed (Participants) | 29 | 30 | 131
  Tailored Prophylaxis | 5417.9 [4683.4 to 6303.9] | 4989.7 [4293.8 to 5842.4] | 4359.8 [3993.8 to 5630.3]
  Weekly Prophylaxis: number analyzed (Participants) | 0 | 0 | 34
  Weekly Prophylaxis |  |  | 3505.2 [3267.9 to 3639.0]
  Personalized Prophylaxis: number analyzed (Participants) | 2 | 1 | 23
  Personalized Prophylaxis | 5457.1 [4435.0 to 6479.1] | 4572.3 [4572.3 to 4572.3] | 3926.7 [3261.8 to 6194.8]
  Episodic: number analyzed (Participants) | 0 | 0 | 13
  Episodic |  |  | 801.7 [286.2 to 1057.7]

6. Secondary Outcome: Physicians' Global Assessment of Participant's Response to rFVIIIFc Regimen Using a 4-Point Scale
Description: Participants were assessed for response to their rFVIIIFc regimen using following 4-point scale: 1=Excellent:bleeding episodes responded to less than or equal to (<=)usual number of injections/dose of rFVIIIFc or rate of breakthrough bleeding during prophylaxis was <= that usually observed; 2=Effective: most bleeding episodes responded to same number of injections and dose, but some required more injections or higher doses, or there was minor increase in rate of breakthrough; 3=Partially Effective: bleeding episodes most often required more injections and/or higher doses than expected or adequate breakthrough bleeding prevention during prophylaxis required more frequent injections and/or higher doses and 4=Ineffective: routine failure to control hemostasis/hemostatic control require additional agents. Total number of scale responses =total count of scale responses for all participants; multiple responses per participant including those at scheduled and unscheduled visits are counted.
Time Frame: Approximately 5 years
Population: FAS- all participants who received at least 1 dose of rFVIIIFc. Data was summarized by treatment regimen for participants from 997HA301/997HA307/997HA309 combined and study from 8HA02PED per planned analysis. Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Measure: Count of Units; unit: Responses
Units Other Than Participants: Responses
Groups:
- rFVIIIFc (Participants From Study 8HA02PED): Participants received rFVIIIFc IV per assigned treatment regimen as follows: Tailored Prophylaxis(TP): 25 IU/kg-65 IU/kg rFVIIIFc every 3-5 days or 2 times/week at approximately 20 IU/kg to 65 IU/kg rFVIIIFc on Day 1 and 40 IU/kg-65 IU/kg rFVIIIFc on Day 4. Weekly P: rFVIIIFc once weekly at approximately 65 IU/kg. Personalized P: If optimal prophylaxis dosing not achieved using TP/WP, Investigator personalized dosing to meet individual participant's needs (i.e. adding "prevention" dose prior to strenuous activity; targeting FVIII trough level of >3%, if bleeding history and/or activity level requires/dosing less frequently). Episodic (On demand): individual dose of rFVIIIFc based on clinical condition, type and severity of bleeding event and if indicated, FVIII levels (per investigator and Sponsor decision). For participants <12 years of age, weekly and episodic treatment regimens were only available once reached at age of 12 years old.
Arm/Group | rFVIIIFc (Participants From Study 8HA02PED) | rFVIIIFc(Participants From Studies 997HA301/997HA307/997HA309)
Number analyzed (Participants) | 61 | 179
Number analyzed (Responses) | 428 | 1252
Responses
  Excellent | 403 | 1061
  Effective | 24 | 186
  Partially Effective | 1 | 5
  Ineffective | 0 | 0

7. Secondary Outcome: Participant's Assessment of Response (Excellent or Good Response) to rFVIIIFc Injections for the Treatment of Bleeding Episodes Using a 4-Point Scale
Description: Using eDiary, participant received rating for treatment response to any bleeding episode (BE) using 4-point scale- 1=Excellent: Abrupt pain relief and/or improvement in signs of bleeding within approximately (approx.) 8 hours (h) after initial injection (inj.); 2=Good: Definite pain relief and/or improvement in signs of bleeding within approx. 8h after an injection, but possibly requiring more than 1 injection after 24-48h for complete resolution; 3=Moderate: Probable/slight beneficial effect within 8h after initial injection and requires more than 1 injection and 4=None: No improvement, or condition worsens within approx. 8h after initial injection. This assessment was to be made approx. 8 to 12h from time the injection was given to treat BE and prior to any additional doses of rFVIIIFc given for same bleeding episode. Percentages are based on the number of bleeding episodes for which a response (excellent or good) was provided for the first injection during the efficacy period.
Time Frame: Approximately 5 years
Population: FAS was analyzed.Data was summarized by treatment regimen for participants from 997HA301/997HA307/997HA309 combined and by age cohort (<6 years and 6 to<12 years old) and treatment regimen for participants from 8HA02PED per planned analysis.Participants were included in summary of more than 1 treatment regimen if their regimen changed during study.
Measure: Count of Units; unit: Injections
Units Other Than Participants: Injections
Arm/Group | rFVIIIFc (8HA02PED [<6 Years Old Age Cohort]) | rFVIIIFc (8HA02PED [6 to <12 Years Old Age Cohort]) | rFVIIIFc[Participants From Studies 997HA301/997HA307/997HA309]
Number analyzed (Participants) | 30 | 31 | 179
Number analyzed (Injections) | 167 | 172 | 1734
Injections
  Tailored Prophylaxis: number analyzed (Injections) | 158 | 171 | 638
  Tailored Prophylaxis | 139 | 155 | 475
  Weekly Prophylaxis: number analyzed (Injections) | 0 | 0 | 341
  Weekly Prophylaxis |  |  | 260
  Personalized Prophylaxis: number analyzed (Injections) | 9 | 1 | 387
  Personalized Prophylaxis | 9 | 1 | 318
  Episodic: number analyzed (Injections) | 0 | 0 | 368
  Episodic |  |  | 338

ADVERSE EVENTS:
Time Frame: From signing Informed Consent Form (ICF) through follow-up (approximately 5 years)
Description: Adverse events (AEs) data was planned to be reported for each group and for the overall participants. AEs emergent during major surgical/rehabilitation periods are analyzed separately as per planned analysis and are presented as separate groups.
Groups:
- rFVIIIFc(Participants From Studies 997HA301/997HA307/997HA309): Participants received rFVIIIFc IV as per their assigned treatment regimen as follows: Tailored Prophylaxis (TP): 25 international unit per kilogram (IU/kg)-65 IU/kg rFVIIIFc every 3-5 days or 2 times/week at approximately 20 IU/kg to 65 IU/kg rFVIIIFc on Day 1 and 40 IU/kg-65 IU/kg rFVIIIFc on Day 4. Weekly P: rFVIIIFc once weekly at approximately 65 IU/kg. Personalized P: If optimal prophylaxis dosing not achieved using TP/WP, Investigator personalized dosing to meet individual participant's needs (options: adding "prevention" dose prior to strenuous activity; targeting FVIII trough level of greater than (>)3 percent (%), if bleeding history and/or activity level requires/dosing less frequently. Episodic (On demand): individual dose of rFVIIIFc IV based on clinical condition, type and severity of bleeding event and if indicated, FVIII levels (per investigator and Sponsor decision). The rate of administration determined by participant's comfort level.
- Overall(Participants From 8HA02PED/997HA301/997HA307/997HA309): All participants who received rFVIIIFc drug in study 8HA01EXT, from studies 8HA02PED and 97HA301/997HA307/997HA309. AEs emergent during major surgical/rehabilitation periods are excluded and are presented as separate groups.
- Participants From Study 8HA02PED- Surgery Subgroup; Participants From 997HA301/997HA307/997HA309- Surgery Subgroup: Participants who required emergent or elective surgery while participating in this study and treated with the dose and regimen of rFVIIIFc as appropriate for the type of surgery. Participants returned to a regular rFVIIIFc regimen once all dosing for the postoperative rehabilitation period had been completed.
Arm/Group | rFVIIIFc (Participants From Study 8HA02PED) | rFVIIIFc(Participants From Studies 997HA301/997HA307/997HA309) | Overall(Participants From 8HA02PED/997HA301/997HA307/997HA309) | Participants From Study 8HA02PED- Surgery Subgroup | Participants From 997HA301/997HA307/997HA309- Surgery Subgroup
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/179 | 0/240 | 0/2 | 0/26
Serious Adverse Events (participants affected / at risk) | 20/61 | 43/179 | 63/240 | 0/2 | 1/26
Other Adverse Events (participants affected / at risk) | 49/61 | 110/179 | 159/240 | 0/2 | 4/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rFVIIIFc (Participants From Study 8HA02PED) (N=61) | rFVIIIFc(Participants From Studies 997HA301/997HA307/997HA309) (N=179) | Overall(Participants From 8HA02PED/997HA301/997HA307/997HA309) (N=240) | Participants From Study 8HA02PED- Surgery Subgroup (N=2) | Participants From 997HA301/997HA307/997HA309- Surgery Subgroup (N=26)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Device breakage (General disorders) | 1 | 0 | 1 | 0 | 0
Device dislocation (General disorders) | 0 | 1 | 1 | 0 | 0
Infusion site mass (General disorders) | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Hepatitis c (Infections and infestations) | 0 | 2 | 2 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Pericoronitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 0 | 6 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 6 | 1 | 7 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Transplant failure (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 1 | 0 | 0
Nuclear magnetic resonance imaging abnormal (Investigations) | 1 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5 | 0 | 0
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 11 | 11 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Bone graft (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Carpal tunnel decompression (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Central venous catheter removal (Surgical and medical procedures) | 4 | 0 | 4 | 0 | 0
Central venous catheterisation (Surgical and medical procedures) | 2 | 1 | 3 | 0 | 0
Circumcision (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Joint arthroplasty (Surgical and medical procedures) | 0 | 1 | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 2 | 2 | 0 | 0
Bleeding varicose vein (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Superior vena caval stenosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rFVIIIFc (Participants From Study 8HA02PED) (N=61) | rFVIIIFc(Participants From Studies 997HA301/997HA307/997HA309) (N=179) | Overall(Participants From 8HA02PED/997HA301/997HA307/997HA309) (N=240) | Participants From Study 8HA02PED- Surgery Subgroup (N=2) | Participants From 997HA301/997HA307/997HA309- Surgery Subgroup (N=26)
Diarrhoea (Gastrointestinal disorders) | 5 | 16 | 21 | 0 | 0
Vomiting (Gastrointestinal disorders) | 8 | 6 | 14 | 0 | 0
Pyrexia (General disorders) | 6 | 5 | 11 | 0 | 0
Seasonal allergy (Immune system disorders) | 9 | 5 | 14 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 6 | 2 | 8 | 0 | 0
Influenza (Infections and infestations) | 3 | 14 | 17 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 37 | 43 | 0 | 0
Pharyngitis (Infections and infestations) | 4 | 2 | 6 | 0 | 0
Tonsillitis (Infections and infestations) | 12 | 2 | 14 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 13 | 19 | 32 | 0 | 0
Viral infection (Infections and infestations) | 4 | 3 | 7 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 7 | 0 | 7 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 11 | 14 | 25 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 15 | 16 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 4 | 10 | 14 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 20 | 27 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 11 | 16 | 0 | 0
Headache (Nervous system disorders) | 10 | 15 | 25 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 17 | 0 | 0
Hypertension (Vascular disorders) | 0 | 9 | 9 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2013-08-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT01454739/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/39/NCT01454739/SAP_001.pdf